CLINICAL TRIAL: NCT02808013
Title: Prospective Randomized, Double-Blind, Placebo Controlled Study of NDS-446 (500 mg/Cap) in Men 45 Years of Age or Older With Moderate to Severe Lower Urinary Tract Symptoms (LUTS)
Brief Title: Study to Evaluate Efficacy and Safety of NDS-446 in Men With Lower Urinary Tract Symptoms (LUTS)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Naturex-Dbs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NDB 2015-001
Record Dates: First submitted 2016-05-31; First posted 2016-06-21 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Lower Urinary Tract Symptoms
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- NDS-446 (Experimental): NDS-446
  Interventions: Drug: NDS-446
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NDS-446
  Arms: NDS-446
Drug: Placebo
  Arms: Placebo

SUMMARY:
Prospective, Randomized, Double-Blind, Placebo Controlled clinical trial to study the efficacy and the safety of NDS-446 (500 mg/cap) in Men 45 years of age or older with moderate to severe lower urinary tract symptoms (LUTS)

ELIGIBILITY:
Inclusion Criteria:

1. Men ≥45 years of age.
2. LUTS, based on IPSS total score ≥8 and <25
3. Peak urinary flow rate (Qmax) ≥4 and ≤15 mL/sec at screening
4. Post Void Residual (PVR) urine volume ≤ 200 mL at screening
5. PSA level at screening < 10 ng/mL. Subjects with a PSA > 4ng/mL and < 10 ng/mL are eligible only if prostate cancer has been ruled out
6. Subjects who understand and speak English
7. Able and willing to give informed consent and comply with all study protocol procedures (diaries and other study tools).

Exclusion Criteria:

1. Not suitable for medical intervention (e.g., requiring TURP, etc.)
2. History of interstitial cystitis, bladder stones, urethral stricture, current prostatitis, acute urinary retention requiring catheterization in the last 3 months, or any other condition suspected to be the cause of LUTS other than BPH
3. Screening serum Creatinine (Cr) or liver function tests [ALT (SGPT), AST (SGOT)] > 3 times the upper limit of normal (ULN) confirmed on a second measurement.
4. Cancer of the prostate or bladder by history or current diagnosis.
5. Prostate nodule(s) on screening digital rectal exam (DRE).
6. Prior surgical procedure of the urinary tract such as TURP, laser prostatectomy, photovaporization of the prostate
7. No minimally invasive surgery to the prostate such as TUMT or TUNA within the last 6 months.
8. Active urinary tract infection.
9. Unstable or uncontrolled medical or psychiatric condition.
10. Abnormal screening labs > 2 times the upper limit of normal (ULN) [for all parameters other than those listed for exclusion criteria#3]
11. Myocardial infarction or CVA within the past 90 days.
12. Requiring ongoing administration of antibiotics, antifungals, antiviral, chemotherapy, steroidal or immunosuppressive treatments.
13. Requiring chronic administration of aspirin at a dose >81 mg/day.
14. Known hypersensitivity to study drug ingredient(s) or allergy to berries.
15. Use of the following medications: alpha blockers (28 days of screening), herbal or nutritional BPH supplements (28 days of screening), OAB medications (28 days of screening), 5 alpha reductase inhibitors (175 days of screening), PDE5 inhibitors (permitted as needed for erectile dysfunction only, but not to exceed 1 dose per week and not to be dosed within 5 days of a visit)
16. Use of an investigational agent (drug, biologic, device, etc.) within 30 days of screening
17. Any reason or condition that in the judgment of the Clinical Investigator(s) may put the subject at unacceptable risk or that may preclude the subject from understanding or complying with the study's requirements.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Change in total IPSS score between baseline and 6 months | 6-month

SECONDARY OUTCOMES:
Change in IPSS subscores (Storage, Voiding, Quality of Life) between baseline and 6 months | 6-month
Change in Patient Global Impression of Improvement/Severity Score (PGIS) between baseline and 6 months | 6-month
Uroflowmetry (Qmax: maximum urinary flow rate, mL/sec) | 6-month
Uroflowmetry (PVR: Post Void Residual Volume, mL) | 6-month
Uroflowmetry (Vol: Volume of urine voided, mL) | 6-month
Sexual performance (SHIM: Sexual Health Inventory for Men) | 6-month
Blood and urine laboratory analysis and incidence of treatment emergent adverse events [Safety and Tolerability] | 6-month
  Blood samples will be collected to measure:
  Prostate Specific Antigen (PSA) Hematology: CBC (complete blood count), differential; reticulocyte count, platelets Serum Chemistries: BUN (blood urea nitrogen), Creatinine, Fasting Blood Glucose, Uric acid, AST (aspartate aminotransferase), ALT (alanine aminotransferase), ALP (alkaline phosphatase), LDH (lactate dehydrogenase), Total and Direct Bilirubin; Total Protein, Albumin, Calcium, Magnesium, Cholesterol, Triglycerides Coagulation: PT (prothrombin time) /PTT (partial thromboplastin time)/ INR (International Normalized Ratio)
  Urine samples will be collected to measure:
  Urinalysis: Urine Protein, Glucose, Microscopic for RBCs (Red blood cell counts), WBCs (white blood cell counts)
  Assessment of adverse events: collection of adverse events on a diary and spontaneously reported adverse events (either via phone calls to the site or during the visits)